CLINICAL TRIAL: NCT01644721
Title: A Two-site Randomised Trial of an Additional Measles Vaccine at 4 Months of Age to Reduce Child Mortality in Rural Areas of Burkina Faso and Guinea-Bissau
Brief Title: Trial of Additional Measles Vaccine to Reduce Child Mortality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Navrongo Health Research Centre, Ghana (Other); Heidelberg University (Other); National Institute for Public Health and the Environment, RIVM, Holland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPTIMUNISE_BHP_early MV
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Measles Vaccine
Keywords: Child mortality; Measles vaccine; Non-specific effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early measles vaccine (Experimental): An additional measles vaccine at 4 months of age, at least 28 days after the third dose of pentavalent vaccine
  Interventions: Biological: Early measles vaccine
- Control (No Intervention): Follows the normal vaccination schedule

INTERVENTIONS:
Biological: Early measles vaccine — Standard Edmonston-Zagreb measles vaccine
  Arms: Early measles vaccine

SUMMARY:
Background: All observational studies and a few randomised controlled trials (RCT) suggest that early measles vaccine (MV), in particular an early two-dose strategy, has a much better effect on overall mortality than later MV. These results suggest that MV has a non-measles related beneficial effect on child survival.

Objective: To evaluate in a two-site RCT the effect on child survival and other health indicators of a two-dose measles vaccination schedule by providing an additional dose of Edmonston-Zagreb (EZ) MV as soon as possible after 4 months of age as well as the standard measles vaccine at 9 months of age. The trials are planned in Guinea-Bissau and Burkina Faso. The investigators will test a 40-43% reduction of mortality at each site separately and a 32% reduction overall. Based on the results from the RCT, the investigators will assess the cost-effectiveness of the intervention.

Design, Guinea-Bissau: Newborns are followed through the Health and Demographic Surveillance System (HDSS) of the Bandim Health Project. Information on routine and campaign vaccinations will be collected regularly through home visits and health centre registers. Four weeks after having received the third dose of pentavalent vaccine (Penta3), the children will be eligible for enrollment in the trial if they are not severely ill. Eligible children will be invited to take part in the trial. Provided parental informed consent is given, the children will be randomised to MV at 4 and 9 months of age or only at 9 months. Cost estimates will be based on consumption of services and average cost per unit. The incremental cost effectiveness ratio will be calculated.

Sample size, follow-up and analyses: To detect a 40% reduction in overall mortality at each site the investigators intend to enroll at least 3,750 children in Guinea-Bissau. The children will be followed for survival and hospitalisations to 3 years of age or to the end of the study after three years. The investigators will analyse the effects by site and combined; by sex and season; possible interactions with other interventions like campaigns with drugs, vaccines or micronutrients will be explored.

Antibody study: 450 children will be enrolled in a subgroup study to examine the effect of maternal antibody levels on subsequent antibody responses to MV. The children will be followed to 24 months of age and samples collected at 4, 9 and 24 months of age.

ELIGIBILITY:
Inclusion Criteria:

Children who

* received the third dose of pentavalent vaccine at least 28 days before enrolment
* are between 4 and 6 months old
* belong to households of the existing HDSS

Exclusion Criteria:

Children

* with serious malformation
* who are severely sick (needing hospitalisation)
* with high fever (>38.5 C axillary temperature)
* who are severely malnourished (mid-upper-arm-circumference (MUAC) < 110 mm and/or bilateral peripheral oedema)
* who have received neonatal vitamin A supplementation
* whose parents/guardians state that they intend to permanently move out of the study area before the child reaches 9 months of age

Ages: 4 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3750 (Actual)
Dates: Start 2012-07; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mortality | 4 months - 3 years
  Overall mortality from 4 months to 3 years by sex and age at enrolment

SECONDARY OUTCOMES:
Mortality | 4 to 9 months of age and from 9 months to 3 years of age
  Mortality from 4 to 9 months of age and from 9 months to 3 years of age
Morbidity | 4 months - 3 years of age
  Hospital admissions, consultations, specific morbidity and measles infection
Growth
Antibody titres

OTHER OUTCOMES:
Immunological markers
  Provided funding becomes available

CONTACTS AND LOCATIONS:
Overall Officials: Cesario Martins, MD,PhD, Principal Investigator — Bandim Health Project; Amabelia Rodrigues, DMSc, Principal Investigator — Bandim Health Project; Peter Aaby, DMSc, Study Director — Bandim Health Project
Locations (1):
- Bandim Health Project, Bissau, Guinea-Bissau

REFERENCES:
- [Background] Aaby P, Martins CL, Garly ML, Bale C, Andersen A, Rodrigues A, Ravn H, Lisse IM, Benn CS, Whittle HC. Non-specific effects of standard measles vaccine at 4.5 and 9 months of age on childhood mortality: randomised controlled trial. BMJ. 2010 Nov 30;341:c6495. doi: 10.1136/bmj.c6495. PMID 21118875
- [Result] Steiniche MM, Thysen SM, Jensen AKG, Rodrigues A, Martins C, Meyrowitsch DW, Aaby P, Fisker AB. The effect of early measles vaccination on morbidity and growth: A randomised trial from Guinea-Bissau. Vaccine. 2020 Mar 4;38(11):2487-2494. doi: 10.1016/j.vaccine.2020.01.096. Epub 2020 Feb 13. PMID 32061387
- [Result] Fisker AB, Nebie E, Schoeps A, Martins C, Rodrigues A, Zakane A, Kagone M, Byberg S, Thysen SM, Tiendrebeogo J, Coulibaly B, Sankoh O, Becher H, Whittle HC, van der Klis FRM, Benn CS, Sie A, Muller O, Aaby P. A Two-Center Randomized Trial of an Additional Early Dose of Measles Vaccine: Effects on Mortality and Measles Antibody Levels. Clin Infect Dis. 2018 May 2;66(10):1573-1580. doi: 10.1093/cid/cix1033. PMID 29177407
- [Derived] Schoeps A, Nebie E, Fisker AB, Sie A, Zakane A, Muller O, Aaby P, Becher H. No effect of an additional early dose of measles vaccine on hospitalization or mortality in children: A randomized controlled trial. Vaccine. 2018 Apr 5;36(15):1965-1971. doi: 10.1016/j.vaccine.2018.02.104. Epub 2018 Mar 6. PMID 29523450